CLINICAL TRIAL: NCT02547064
Title: Stylet Angulation of Seventy Degrees Reduced Time to Intubation With the GlideScope®: A Prospective Randomized Trial
Brief Title: Effect of Modified Stylet Angulation on the Intubation With GlideScope®
Acronym: GlideMStylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GlideMStylet
Record Dates: First submitted 2015-09-01; First posted 2015-09-11 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Cholecystitis; Stomach Cancer
Keywords: intubation; stylet; videolaryngoscope
MeSH Terms: conditions — Cholecystitis; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 90 degree (Active Comparator): The ETT with the 90° angle stylet was bent at a point 8 cm from its distal end.
  Interventions: Procedure: Glidescope guided intubation; Device: GlideScope®
- 70 degree (Experimental): The ETT was bent by 70° at a point 6 cm from its distal end and the proximal portion of the ETT was formed as the shape of the GL blade until the point of the handle.
  Interventions: Procedure: Glidescope guided intubation; Device: GlideScope®

INTERVENTIONS:
Procedure: Glidescope guided intubation
Device: GlideScope®

SUMMARY:
The GlideScope® videolaryngoscope usually visualize glottis better than the conventional laryngoscope. Under the visualization of glottis by GlideScope®, the insertion of endotracheal tube, however, is challenging.

The goal of this study was to determine which of two stylet (70° vs 90°) was better, as determined by time to intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring endotracheal intubation for general anesthesia

Exclusion Criteria:

* Difficult airway
* Rapid sequence induction
* Recent sore throat
* Fragile teeth
* Contraindication for videolaryngoscope
* Head and neck surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

REFERENCES:
- [Derived] Lee YC, Lee J, Son JD, Lee JY, Kim HC. Stylet angulation of 70 degrees reduces the time to intubation with the GlideScope(R): A prospective randomised trial. J Int Med Res. 2018 Apr;46(4):1428-1438. doi: 10.1177/0300060517741065. Epub 2018 Jan 14. PMID 29332445

RESULTS

PARTICIPANT FLOW:
Groups:
- 90 Degree: The ETT with the 90° angle stylet was bent at a point 8 cm from its distal end.
  Glidescope guided intubation
  GlideScope®
- 70 Degree: The ETT was bent by 70° at a point 6 cm from its distal end and the proximal portion of the ETT was formed as the shape of the GL blade until the point of the handle.
  Glidescope guided intubation
  GlideScope®
Period: Overall Study
Arm/Group | 90 Degree | 70 Degree
Started | 81 | 81
Completed | 78 | 79
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 90 Degree | 70 Degree | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 79 | 157
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 57 (16) | 58 (14)
Sex/Gender, Customized [Number; unit: participants]
  Female | 37 | 33 | 70
  Male | 41 | 46 | 87
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 78 | 79 | 157

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: Time from the insertion of the Glidescope blade to the measurement of end tidal CO2 (>30 mmHg)
Time Frame: Intraoperative intubation
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
sec | 47.2 (35.8) | 31.0 (17.5)

2. Secondary Outcome: Success Rate of Intubation
Description: The number of patients in which the intubation was successful at the first time.
Time Frame: Intraoperative intubation
Measure: Count of Participants; unit: Participants
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
Participants | 68 | 79

3. Secondary Outcome: Difficulty of Intubation Measured Using Visual Analogue Scale
Description: Difficulty of intubation will be measured using visual analogue scale (0:easiest, 100:most difficult).
Time Frame: Intraoperative intubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
units on a scale | 35 (29) | 22 (24)

4. Secondary Outcome: Number of Participants for Whom External Laryngeal Manipulation Was Necessary
Description: External laryngeal manipulation is defined as the compression of neck for the facilitation of laryngeal view. Number of participants for whom external laryngeal manipulation was necessary will be measured.
Time Frame: Intraoperative intubation
Measure: Count of Participants; unit: Participants
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
Participants | 14 | 3

5. Secondary Outcome: Cormack-Lehan Grade
Description: The grade of Cormack-Lehan was assessed as I/II/III/IV (I: Full view of glottis, II: Partial view of glottis, III: Only epiglottis seen, none of glottis seen, IV: Neither glottis nor epiglottis seen). Grade I was considered better outcomes.
Time Frame: Intraoperative intubation
Measure: Count of Participants; unit: Participants
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
Participants
  I | 70 | 68
  II | 7 | 9
  III | 1 | 2
  IV | 0 | 0

6. Secondary Outcome: Mallampati Grade
Description: The Mallapati grade was assessed as I/II/III/IV (I: Soft palate, uvula, fauces, pillars visible, II: Soft palate, uvula, fauces visible, III: Soft palate, base of uvula visible, IV: Only hard palate visible). Grade I was considered better outcomes.
Time Frame: Intraoperative anesthetic induction
Measure: Count of Participants; unit: Participants
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
Participants
  I | 36 | 32
  II | 25 | 33
  III | 10 | 8
  IV | 7 | 6

7. Secondary Outcome: Thyromental Distance
Description: The thyromental distance was measured.
Time Frame: Intraoperative anesthetic induction
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
mm | 79.1 (23.6) | 78.5 (24.5)

8. Secondary Outcome: Postoperative Sore Throat Measured Using Visual Analogue Scale
Description: Postoperative sore throat will be measured using visual analogue scale (0:no pain, 100: worst pain imaginable)
Time Frame: at 1, 24 hr postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
units on a scale
  1 h postoperatively | 16 (27) | 13 (25)
  24 h postoperatively | 10 (20) | 8 (18)

9. Secondary Outcome: Mean Blood Pressure
Description: Mean blood pressure is measured before and 2 min after intubation.
Time Frame: Intraoperative intubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
mmHg
  Before intubation | 77 (12) | 78 (14)
  2 min after intubation | 105 (22) | 108 (25)

10. Secondary Outcome: Heart Rate
Description: Heart rates are measured before and 2 min after intubation.
Time Frame: Intraoperative intubation
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
beats per minute
  Before intubation | 73 (15) | 73 (17)
  2 min after intubation | 93 (19) | 93 (16)

11. Secondary Outcome: Airway Injury
Description: Larynx injury is assessed.
Time Frame: Intraoperative intubation
Measure: Count of Participants; unit: Participants
Arm/Group | 90 Degree | 70 Degree
Number analyzed (Participants) | 78 | 79
Participants | 5 | 0

ADVERSE EVENTS:
Arm/Group | 90 Degree | 70 Degree
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 0/78 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No